CLINICAL TRIAL: NCT05214950
Title: A Randomized Controlled Trial of the Effect of Oxygen Reserve Index Monitoring for Preventing Hypoxia in Pediatric Airway Surgery
Brief Title: Oxygen Reserve Index in Airway Surgery in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2112-055-1281
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Hypoxemia During Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ORI monitoring (Experimental): SpO2, ECG, NIBP, and oxygen reserve index monitoring
  Interventions: Device: ORI monitoring
- Standard monitoring (No Intervention): SpO2, ECG, NIBP monitoring

INTERVENTIONS:
Device: ORI monitoring — Oxygen reserve index monitoring during the surgery
  Arms: ORI monitoring

SUMMARY:
This study aimed to identify the effect of oxygen reserve index monitoring on the occurrence of oxygen desaturation (<90%) in pediatric patients undergoing airway surgery.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients receiving airway surgery

Exclusion Criteria:

* baseline oxygen saturation less than 95%
* patients diagnosed as respiratory distress syndrome, bronchopulmonary dysplasia, pneumonia requiring oxygen supplements

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | from induction of anesthesia to end of operation, about 3 hours
  Oxygen desaturation <= 90%

SECONDARY OUTCOMES:
Hypoxemia duration | from induction of anesthesia to end of operation, about 3 hours
  Total length of time patient experienced hypoxemia during hypoxemic event (oxygen desaturation <= 90%)
Incidence and duration of severe hypoxemia | from induction of anesthesia to end of operation, about 3 hours
  incidence and duration of oxygen desaturation <=85%
Rescue oxygenation | from induction of anesthesia to end of operation, about 3 hours
  the number of the surgical procedure is interrupted and the anesthetist attempts to improve oxygenation of the child.
Hemodynamic instability | from induction of anesthesia to end of operation, about 3 hours
  occurrence of hypotension requiring treatment, bradycardia requiring treatment, cardiac arrest with or without return of spontaneous circulation at any time during procedure
unexpected pediatric intensive care admission | from induction of anesthesia to end of operation, about 3 hours
  requirements of unexpected pediatric intensive care admission
unanticipated postoperative mechanical support | from induction of anesthesia to end of operation, about 3 hours
  Requirement for unanticipated postoperative mechanical ventilation or any other form of non-invasive ventilation including high-flow nasal oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided